CLINICAL TRIAL: NCT03418480
Title: Therapeutic HPV Vaccine (BNT113) Trial in HPV16 Driven Carcinoma
Brief Title: HARE-40: HPV Anti-CD40 RNA vaccinE
Acronym: HARE-40
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of Southampton (Other)
Collaborators: BioNTech SE (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RHMCAN0983; 2014-002061-30 (EudraCT Number); ISRCTN51789191 (Other: ISRCTN Reference No.)
Record Dates: First submitted 2017-11-15; First posted 2018-02-01 (Actual); Last update posted 2024-02-07 (Actual); Status verified 2024-02

CONDITIONS: Human Papilloma Virus Related Carcinoma; Head and Neck Neoplasm; Cervical Neoplasm; Penile Neoplasms Malignant; Unknown Primary Tumors
MeSH Terms: conditions — Head and Neck Neoplasms; Uterine Cervical Neoplasms; Penile Neoplasms; Neoplasms, Unknown Primary

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- RNA Vaccine A (Experimental): Arm 1A: 15 (6+9) patients with previously treated HPV16+ head and neck squamous cell carcinoma receiving increasing doses of HPV vaccine.
  - COMPLETE no longer recruiting
  Interventions: Drug: BNT113
- RAN Vaccine B (Experimental): Arm 1B: 29 (15+14) patients with HPV16+ advanced disease receiving increasing doses of HPV vaccine.
  OPEN to recruitment
  Interventions: Drug: BNT113

INTERVENTIONS:
Drug: BNT113 — Intradermal vaccine

SUMMARY:
HARE-40 is a phase I/II vaccine dose escalation study with two different arms: Arm 1A will perform intrapatient dose escalation in patients with previously treated HPV16+ Head & Neck Cancer using two dose cohorts to establish a safe, tolerable and recommended dose of HPV vaccine.

Arm 1B will perform intrapatient dose escalation in patients with advanced HPV16+ cancer (head and neck, anogenital, penile, cervical and other) using a single cohort to establish a safe, tolerable and recommended dose of HPV vaccine.

DETAILED DESCRIPTION:
HARE-40 is a phase I/II vaccine dose escalation trial with two arms (Arm 1A and Arm 1B) in which we will test BNT113 as monotherapy. We will undertake a multi-centre phase I, open label trial in patients with previous HPV16+ HNSCC without current clinical evidence of disease (Arm 1A) and in patients with HPV16+ advanced disease (Arm 1B). The HPV16 antigen-specific immune response will be evaluated before and after treatment in circulating blood and, where samples have been collected, in tumour and skin biopsies.

Arms 1A and 1B will escalate BNT113 in each patient (intrapatient dose escalation) up to the specified target dose of the cohort to establish a safe, tolerable and recommended dose of BNT113 in patents who are disease free (Arm 1A) and those with advanced disease (Arm 1B).

Subset of patients in Arm 1B will also be assessed for response to the vaccine in terms of a significant increase of immune cells following BNT113 administration and according to irRECIST1.1 (all 29 patients including the expansion cohort) and other endpoints.

ELIGIBILITY:
Inclusion Criteria:

Arm 1A:

* Previous HPV16+ head and neck squamous cell carcinoma.
* At least 12 months after completion of treatment.
* Within 5 years of treatment completion.
* Currently no clinical evidence of disease.
* ECOG performance status 0 or 1.

Arm 1B:

* HPV16+ head and neck, cervical, anogenital and penile carcinoma patients with recurrent disease.
* Intention to treat is palliative.
* Patient willing to have repeated tumour biopsies and re-biopsy deemed safe and feasible clinically.
* Tissue samples available confirming HPV16+ disease to send to Central Laboratory.

Exclusion Criteria:

* Patients unable to consent.
* Any patient who has been previously vaccinated in any Arm of the trial.
* <18 years
* Systemic steroids (prednisolone >10 mg/day or equivalent) or other drugs with a likely effect on immune competence are forbidden during the trial. The predictable need of their use will preclude the patient from trial entry. Replacement steroids for adrenal insufficiency/failure are allowed.
* Major surgery in the preceding three to four weeks, which the patient has not yet recovered from.
* Patients who are of high medical risk because of non-malignant systemic disease, as well as those with active uncontrolled infection.
* Patients with clinically relevant autoimmune disease will be excluded.
* Patients who are known to be allergic to any of the excipients or constituents of the vaccine
* Patients with any other condition which in the Investigator's opinion would not make the patient a good candidate for the clinical trial, such as concurrent congestive heart failure or prior history of New York Heart Association (NYHA) class III/IV cardiac disease.
* Current malignancies at other sites, with the exception of adequately treated basal or squamous cell carcinoma of the skin. Cancer survivors, who have undergone potentially curative therapy for a prior malignancy, have no evidence of that disease for five years and are deemed at low risk for recurrence, are eligible for the study.
* Patients who are serologically positive for or are known to suffer from Hepatitis B, C, Syphilis or HIV. Counselling will be offered to all patients prior to testing.
* Patients who have a positive pregnancy test or who are breast feeding.
* Fertile males or females who are unable or unwilling to use an effective method of birth control (eg. condom with spermicide, diaphragm with spermicide, birth control pills, injections, patches, intrauterine device, or intrauterine hormone-releasing system) during study treatment and until 28 days after patients finish the study treatment.
* Elevated Liver Function Tests - ALT >3.0 x ULN, AST >3.0 x ULN, Bilirubin >3.0 x ULN.
* Any other investigational drug within 28 days or 5 half-lives depending on what gives the longer range before the first treatment of this study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2017-04-11 (Actual); Primary Completion 2023-11-01 (Actual); Study Completion 2024-01-24 (Actual)

PRIMARY OUTCOMES:
Dose Limiting Toxicity (DLT) according to CTCAE version 4.03 (Arm 1A) | 3 months
  Safe and tolerable dose of clinically disease free patients (Arm 1A) - Determination of a suitable dose of HPV RNA

CONTACTS AND LOCATIONS:
Overall Officials: Christian Ottensmeier, Prof, Study Chair — University of Liverpool; Ioannis Karydis, Dr, Principal Investigator — University Hospitals Southampton NHS Foundation Trust
Locations (2):
- United Kingdom (2):
  - Univeristy Hospitals Southampton NHS Foundation Trust, Southampton, Hampshire
  - The Christie NHS Foundation Trust, Manchester

IPD SHARING:
Plan to Share IPD: No